CLINICAL TRIAL: NCT03062709
Title: Urine Cotinine in Children and Parental Behavior Modification: A Pilot Study
Brief Title: A Study of Tobacco Smoke and Children With Respiratory Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Deirdre Burns, Principal Investigator, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 986404-3
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Bronchiolitis; Pneumonia; Reactive Airway Disease; Asthma; Tobacco Smoking; Tobacco Cessation; Bronchopulmonary Dysplasia
Keywords: tobacco cessation; bronchiolitis; pneumonia; pediatric; environmental tobacco smoke; secondhand tobacco smoke; thirdhand tobacco smoke; tobacco smoke; asthma; reactive airway disease; bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchiolitis; Pneumonia; Pulmonary Disease, Chronic Obstructive; Asthma; Tobacco Smoking; Tobacco Use Cessation; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Breathe Easy Coalition written materials provided to parent/guardian, plus Maine Tobacco Helpline referral provided to smoking adult in the home, plus testing of the child's urine cotinine and results reported to parent/guardian
  Interventions: Behavioral: Breathe Easy Coalition written materials; Behavioral: Maine Tobacco Helpline; Diagnostic Test: Urine cotinine testing

INTERVENTIONS:
Behavioral: Breathe Easy Coalition written materials — written materials about secondhand and thirdhand environmental smoke exposure in children
Behavioral: Maine Tobacco Helpline — referral to tobacco cessation counselor, helpline calls adult referred to provide counseling over the phone.
Diagnostic Test: Urine cotinine testing — the child's urine is tested for cotinine, which is produced when the body absorbs nicotine. These results are communicated to the child's parent/guardian.

SUMMARY:
This study aims to assess the feasibility of using an intervention for environmental smoke exposure in children that uses cotinine testing results with written materials and telephone counseling for a potential future study of parents whose children are admitted with respiratory illnesses to The Barbara Bush Children's Hospital in Portland, Maine.

DETAILED DESCRIPTION:
Children who are regularly exposed to environmental tobacco smoke (ETS) are at a greater risk for developing respiratory disease. Given the strong relationship between parental smoking and child health, many studies have evaluated the efficacy of interventions to modify parental smoking behavior and thereby reduce children's exposure to second- and thirdhand tobacco smoke, including the use of cotinine levels in children. There are several local ETS exposure intervention programs for The Barbara Bush Children's Hospital patient population and their families. The state of Maine and MaineHealth fund a free 24-hour tobacco cessation hotline (The Maine Tobacco Helpline) which combines evidence-based behavioral counseling techniques and free nicotine replacement therapy (gum, lozenge, or patch). MaineHealth also runs a tobacco cessation campaign (The Breathe Easy Coalition) that provides print materials and trainings aimed to reduce smoking in public housing, hospitals, behavioral health facilities, and higher education. The Breathe Easy Coalition's Smoke-Free Housing program provides education about the effects of secondhand and thirdhand tobacco smoke and asks families to pledge to keep tobacco smoke out of their home. This study aims to combine all three of these strategies (child cotinine feedback, tobacco cessation counseling, and written materials on ETS) to create a cohesive ETS exposure reduction program for the Barbara Bush Children's Hospital inpatient population, and determine the feasibility of a future study that would evaluate whether cotinine testing is helpful for changing smoking behaviors in this target population.

ELIGIBILITY:
Inclusion Criteria:

* age 0 to 10 years old
* admitted to The Barbara Bush Children Hospital for bronchiolitis, pneumonia, bronchopulmonary dysplasia, or asthma
* the child lives with an adult who smokes cigarettes

Exclusion Criteria:

* Non-English-speaking and -reading adults will be excluded as our interventions are in English.
* Children over the age of 10 will be excluded as we wanted to avoid children who themselves smoke, given that we will not have a confidential way to assess this.
* Breastfeeding children will be excluded as nicotine is transferrable in breast milk.
* Families (meaning the parent or guardian, the child, and any smoking coinhabiting caregiver) will be excluded if the parent or the smoking adult is a minor, as they would not be able to give consent for participation.
* Children in foster care or whose guardian is the state will be excluded as we are unlikely to achieve timely consent.
* Families who do not reside in Maine will be excluded as The Maine Tobacco Helpline is not able to provide services for out-of-state residents.
* Children readmitted to the hospital during our study period will be excluded if they have already participated in this study during a previous admission.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of acceptance of a smoking cessation intervention | one month for each patient
  Rate of acceptance of participation in each of the three smoking cessation interventions in this patient population at BBCH--written materials, phone counseling, and urine cotinine testing.

SECONDARY OUTCOMES:
Rate of positive urine cotinine in children admitted with positive tobacco smoke exposure history. | 24 hours for each patient
  We will assess the number of children who have a positive smoke exposure history and whose urine is positive for cotinine.
Staff hours required to provide a smoking cessation intervention | one month for each patient
  The staff hours required to provide timely consent and sample collection, and the staff hours required to collect data and provide test results
Rate of acceptance of follow-up urine cotinine testing | one month for each patient
  Rate of parental acceptance of possible follow-up cotinine testing were it provided in a future study.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Burns, MD, MPH, Principal Investigator — MaineHealth
Locations (1):
- The Barbara Bush Children's Hospital at Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Breathe Easy Coalition — http://breatheeasymaine.org/